CLINICAL TRIAL: NCT07189429
Title: PA-100 Workflow Assessment
Brief Title: Clinical Impact Analysis of PA-100 AST in a Spanish GP Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sysmex Europe GmbH (Industry)
Collaborators: Sysmex España S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SEU-MSD-PA100II
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: UTI - Urinary Tract Infection; UTI - Lower Urinary Tract Infection; AMR; Cystitis Acute; Cystitis Bacterial
Keywords: Clinical impact investigation; PA-100 AST
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients were managed according to local guidelines for uncomplicated community acquired urinary tract infection
- Standard of Care with PA.100 AST (Experimental): Patients were managed according to local guidelines for uncomplicated community acquired urinary tract infection while having the additional information of PA-100 AST available during treatment decision.
  Interventions: Diagnostic Test: PA-100 AST

INTERVENTIONS:
Diagnostic Test: PA-100 AST — Results of the PA-100 AST were made available to the treating physician
  Arms: Standard of Care with PA.100 AST

SUMMARY:
Assessment of workflow implications of the PA-100 AST System.

Using well-defined data collection protocols, the study comprises the following:

* Collection of clean-catch midstream urine samples
* Measurement of specimens on the PA-100 AST System

  o Antibiotics tested: Amoxicillin/clavulanic acid (AMC), Ciprofloxacin (CIP), Trimethoprim (TRI), Fosfomycin (FOS) and Nitrofurantoin (NIT)
* Treatment of patients according to the results of the tests on the PA-100 AST System
* Collection of data about patient treatment and antibiotic prescription when the PA-100 AST System is not used (study baseline)
* Collection of patient related information
* Collection of workflow-related information, including doctors and nurses at the test location
* Evaluation of changes in the prescription behaviour when using the PA-100 AST System, compared to current practice at the Test Location

DETAILED DESCRIPTION:
Uncomplicated cystitis in females is among the most frequent community-acquired infections. Urinary tract infection (UTI) is classified as uncomplicated if it occurs in patients with a structurally and functionally normal urinary tract in otherwise healthy, non-pregnant women. Such acute uncomplicated UTIs occur frequently and are associated with high morbidity. Approximately one third of women up to 24 years of age have experienced uncomplicated UTI.

The current gold standard for UTI diagnosis is urine culture of a midstream, clean-catch urine specimen, followed by antibiotic susceptibility testing (AST). UTI patients are often treated empirically with antibiotics, and most guidelines recommend starting antibiotic treatment without or before urine culture and AST results become available. This results in patient treatment without laboratory evidence or at least in a delay of targeted antibacterial therapy by approximately 48 h, when applicable. Due to the continually changing local rates of antimicrobial resistance, empiric treatments do not ensure appropriate stewardship and can result in therapeutic failure.

Therefore, rapid and accurate diagnosis, leading to evidence-based treatment, is essential to achieve a timely and effective therapy.

With antibiotic resistance rates for common antibiotics reaching values as high as 20% of bacteria, the current empiric treatment at GP level carries the risk of clinical failure and the possibility to further increase the prevalence of antibiotic resistant strains.

A point-of-care test (POCT) is defined as a diagnostic tool applicable near the site of patient care that has the potential to provide an accurate and fast diagnostic result. Several POCTs for UTI have been developed and are currently commercially available to detect the presence of bacteria or their activity in urine samples, including both culture-based and enzymatic assays, also in automated format. Existing POC tests, however, cannot provide rapid AST results during the patients first doctor visit, resulting in a delay of personalized treatment. It is the goal of the PA-100 AST System to perform a fast, automated and objective results for bacteriuria detection and AST results in less than 45 minutes and independent from the operator determination of bacteriuria and AST test.

The following investigation serves as a pilot study to better understand the potential and performance of the PA-100 Analyzer in combination with the PA-AST Panel U-0501. PA-100 AST System refers to PA-100 Analyzer in conjunction with the PA-AST Panel U-0501.

ELIGIBILITY:
Inclusion Criteria:

Patients were recruited according to the following criteria: non-pregnant female, >18 years old, presenting with acute UTI symptoms that had been present for < 7 days (symptoms according to the current guidelines [EAU]), with no antibiotic treatment within the previous 7 days, positive urine dipstick for leukocyte esterase (LEU) and/or nitrites (NIT) and who provided a clean-catch mid-stream urine sample.

Exclusion Criteria:

Withdraw of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Frequency of antibiotic prescription | At initial GP visit

SECONDARY OUTCOMES:
Type of antibiotic prescribed | At initial GP visit

CONTACTS AND LOCATIONS:
Overall Officials: Jose Medina Polo, Principal Investigator — Urología, Hospital 12 de Octubre. Servicio Madrileño de salud
Locations (1):
- Centro de Salud Ensanche de Vallecas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Not included in ethical review assesment